CLINICAL TRIAL: NCT05449236
Title: A Reliability and Validity Study of Urdu Version of Western Ontario And MacMaster Osteoarthritis Index Among Pakistani Primary Knee Osteoarthritis Patients
Brief Title: A Reliability and Validity Study of Urdu Version of Western Ontario And MacMaster Osteoarthritis Index
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00251
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Knee Osteoarthritis
Keywords: Western Ontario And MacMaster Osteoarthritis Index; Urdu Version; Reliability; Validity; Knee Osteoarthritis; Lequesne Index
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to translate and culturally adapt Western Ontario And MacMaster Osteoarthritis Index into Urdu language and to investigate its reliability and validity Pakistani population with primary knee osteoarthritis while assessing its correlation with Lequesne Index.

DETAILED DESCRIPTION:
As per preceding commendation, Western Ontario And MacMaster Osteoarthritis Index will be translated into Urdu language from its English version and adapted culturally in Pakistan. Among primary knee osteoarthritis population, Western Ontario And MacMaster Osteoarthritis Index will be distributed among 87 patients recruited by convenience sampling technique under the pre-defined inclusion and exclusion criteria after signing consents forms. For testing inter-observer reliability and intra-observer reliability of Western Ontario And MacMaster Osteoarthritis Index and Lequesne Index will be administrated by two observers, on the same day, with a time interval of 2 hours between 1st and 2nd conduction. As for the 3rd conduction, it will be carried out after seven days by the first observer, for intra-observer assessment. Statistical Package of Social Sciences software version 24 will be used for the purpose of data entry and analysis. Internal consistency will be assessed by using an intra-class correlation coefficient. The Western Ontario And MacMaster Osteoarthritis Index will be evaluated for content validity, construct validity, criterion validity and responsiveness

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients
* Age above 40 years
* Participants with primary knee Osteoarthritis
* Patients willing to participate.

Exclusion Criteria:

* History or presence of ;
* Rheumatic diseases,severe articulation inflammation and cardiac disease.
* Participants with secondary knee Osteoarthritis.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pakistani population with primary knee Osteoarthritis will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Western Ontario And MacMaster Osteoarthritis Index | 1st day
  Western Ontario And MacMaster Osteoarthritis Index is an instrument which used to check the results of treatment. Western Ontario And MacMaster Osteoarthritis Index is valid and reliable Outcome measure for Pain and Activity of Daily Livings.
Lequesne Index | 1st day
  The Lequesne Index is a 10-question survey given to patients with osteoarthritis of the knee. It has five questions pertaining to pain or discomfort, one question dealing with maximum distance walked, and four questions about activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No